CLINICAL TRIAL: NCT02585440
Title: A Phase 1, Randomized, Partial-Blind, Placebo-controlled, Sequential Dose Group, Ascending, Multiple Dose Study of the Safety, Tolerability and Pharmacokinetics, With Food Effect, of CMX157 in Healthy Subjects
Brief Title: A Multiple Dose Study of the Safety, Tolerability and PK of CMX157 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ContraVir Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: ContraVir (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTRV-CMX-102
Record Dates: First submitted 2015-09-30; First posted 2015-10-23 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Infectious Disease
MeSH Terms: conditions — Communicable Diseases | interventions — hexadecyloxypropyl 9-(2-(phosphonomethoxy)propyl)adenine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group A (Experimental): CMX157, tablet, 5 mg, QD, 14 days versus CMX157 placebo, 5 mg, tablet, QD, 14 days
  Interventions: Drug: CMX157; Drug: placebo
- Group B (Experimental): CMX157, tablet, 10 mg, QD, 14 days versus CMX157, placebo tablet, 10 mg, QD, 14 days
  Interventions: Drug: CMX157; Drug: placebo
- Group C (Experimental): CMX157, tablet, 25 mg, QD, 14 days versus placebo CMX157, placebo tablet, 25 mg, QD, 14 days
  Interventions: Drug: CMX157; Drug: placebo
- Group D (Experimental): CMX157, tablet, 50 mg, QD, 14 days versus CMX157, placebo tablet, 50 mg, QD, 14 days
  Interventions: Drug: CMX157; Drug: placebo
- Group E (Experimental): CMX157, tablet, 100 mg, QD, 14 days versus CMX157, placebo tablet, 100 mg, QD, 14 days
  Interventions: Drug: CMX157; Drug: placebo

INTERVENTIONS:
Drug: CMX157 — Oral tablet
  Other Names: Lipid Conjugate TFV
Drug: placebo — Oral tablet

SUMMARY:
This is a phase 1 study to evaluate the safety and tolerability of multiple oral doses of CMX157 at increasing dose levels.

DETAILED DESCRIPTION:
This is a phase 1 study to evaluate the safety and tolerability of multiple oral doses of CMX157 at increasing dose levels, in a fasted state and a fed state.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-55.
* Capable of giving written informed consent.
* Capable of completing study requirements.

Exclusion Criteria:

* Positive result for HIV, HBV, or HCV.
* History or medical condition which could impact patient safety.
* Current or past abuse of alcohol or illicit drugs.
* Participation in another clinical trial within the past 30 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety and tolerability of multiple oral doses of CMX157 at increasing dose levels. | 28 days
  Capture adverse events, physical examinations, ECGs and clinical laboratory panels.

SECONDARY OUTCOMES:
Evaluation of the pharmacokinetics of multiple doses of oral CMX157 in a fasted state. | 28 days
  Measuring Cmax: the peak plasma concentration.
Evaluation of the pharmacokinetics of multiple doses of oral CMX157 in a fed state. | 28 days
  Measuring Cmax: the peak plasma concentration.
Evaluation of the pharmacokinetics of multiple doses of oral CMX157 in a fasted state. | 28 days
  Measuring Tmax: the time Cmax was observed.
Evaluation of the pharmacokinetics of multiple doses of oral CMX157 in a fed state. | 28 days
  Measuring Tmax: the time Cmax was observed.
Evaluation of the pharmacokinetics of multiple doses of oral CMX157 in a fasted state. | 28 days
  Measuring AUC: area under the plasma concentration versus time curve.
Evaluation of the pharmacokinetics of multiple doses of oral CMX157 in a fed state. | 28 days
  Measuring AUC: area under the plasma concentration versus time curve.
Evaluation of the pharmacokinetics of multiple doses of oral CMX157 in a fasted state. | 28 days
  Measuring Cmin: minimum observed plasma concentration.
Evaluation of the pharmacokinetics of multiple doses of oral CMX157 in a fed state. | 28 days
  Measuring Cmin: minimum observed plasma concentration.

CONTACTS AND LOCATIONS:
Overall Officials: John Sullivan-Bolyai, MD, MPH, Study Chair — ContraVir
Locations (1):
- Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes